CLINICAL TRIAL: NCT00451009
Title: Safety and Effectiveness of Freeze and Thaw Media Kits for the Manufacturing of Oocytes for Future Use in Assisted Reproductive Technology
Brief Title: Safety and Efficacy of Freezing and Thawing of Human Eggs in Assisted Reproductive Technology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: ViaCell (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRH-01
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Infertility
Keywords: IVF; Male factor infertility; Cryopreservation; Cryoprotective agents; Egg Freezing
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Viacell's product Media Kits

SUMMARY:
The purpose of this study is to determine the effectiveness of the ViaCell's product media for freezing and thawing human eggs for future use in assisted reproductive technology.

DETAILED DESCRIPTION:
ViaCell's product is an investigational product intended to broaden reproductive options for women through freezing and thawing of human eggs. The egg is a large cell with a high water content, historically making it difficult to freeze. It uses a choline chloride-based media designed to protect the cells from damage during the freezing process with the goal of making it possible to successfully store and thaw eggs for future use.

Following informed consent, female subjects will be screened according to the inclusion/exclusion criteria of the protocol and eligible subjects will undergo hormonal stimulation using standard IVF drugs.

ELIGIBILITY:
Inclusion Criteria:

* Women 21-35 years of age
* Women with male factor infertility seeking IVF treatment
* Negative history of female infertility
* Non-smoking for at least 1 year

Exclusion Criteria:

* Greater than one miscarriage
* More than one previous failed IVF attempt

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Live birth

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Reproductive Science Center, San Ramon, California
  - South Florida Institute for Reproductive Medicine, South Miami, Florida
  - University of Iowa Hospitals and Clinics, Center for Advanced Reproductive Care, Iowa City, Iowa
  - Boston IVF, Waltham, Massachusetts